CLINICAL TRIAL: NCT07306273
Title: A Single-Arm, Open-Label Clinical Study of Irreversible Electroporation(IRE) Combined With the Dual-Function Antibody PD-1/CTLA-4 (Apalulizumab) for the Treatment of Locally Advanced Pancreatic Cancer Following Failure of First-Line AG Therapy
Brief Title: IRE Combined With the Dual-Function Antibody PD-1/CTLA-4 for the Treatment of LAPC Following Failure of First-Line AG Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhongmin Wang, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-608
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Adenocarcinoma Locally Advanced
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRE Combined with the Dual-Function Antibody PD-1/CTLA-4 (Experimental)
  Interventions: Radiation: Irreversible electroporation; Drug: Dual-Function Antibody PD-1/CTLA-4

INTERVENTIONS:
Radiation: Irreversible electroporation — Irreversible electroporation for pancreatic tumor
Drug: Dual-Function Antibody PD-1/CTLA-4 — Dual-Function Antibody PD-1/CTLA-4 iv. injection

SUMMARY:
The study explores the efficacy and safety of irreversible electroporation(IRE) combined with the dual-function antibody PD-1/CTLA-4 (Apalulizumab) for the treatment of locally advanced pancreatic cancer following failure of first-line AG therapy. This research aims to accumulate more clinical evidence and treatment options for second-line therapy in locally advanced pancreatic cancer following failure of first-line regimen.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above, with no gender restrictions;
* Pathologically confirmed pancreatic cancer (originating from the pancreatic ductal epithelium), with clinical records indicating locally advanced pancreatic cancer;
* Clinical records indicating previous failure of standard AG treatment (having received at least one cycle of standardized chemotherapy, with disease progression or intolerance during treatment, or disease progression after the end of treatment);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
* Adequate organ function, meeting the following criteria:

  a. Hematological tests:
  1. Neutrophils ≥ 1.5 × 10⁹ /L;
  2. White blood cells ≥ 3.0 × 10⁹ /L;
  3. Platelets ≥ 85 × 10⁹ /L;
  4. Hemoglobin ≥ 70 g/L; b. Biochemical tests:

  <!-- -->

  1. Total bilirubin ≤ 2× upper limit of normal (ULN) (for subjects with biliary obstruction, after biliary drainage ≤ 2.5 × ULN);
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) in metastatic subjects ≤ 5 × ULN;
  3. Albumin level ≥ 28 g/L;
  4. Creatinine clearance rate ≥ 60 ml/min; c. Cardiac function tests:

  <!-- -->

  1. Normal electrocardiogram (ECG) or ECG abnormalities deemed clinically insignificant by the investigator;
  2. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal;
* At least 3 weeks post-surgery, radiotherapy, chemotherapy, or other anti-tumor treatments, with general physical condition or related adverse reactions having recovered (toxicity ≤ grade 1) or stabilized;
* Willing to participate and sign the informed consent form;
* Good compliance and agreement to cooperate with survival follow-up.

Exclusion Criteria:

* Metastatic pancreatic cancer or has previously undergone interventional treatment for pancreatic cancer;
* Subjects with ascites requiring clinical intervention (including moderate to large amounts of ascites; subjects with ascites need to be stable for more than 4 weeks after drainage);
* Clinically severe gastrointestinal diseases (including bleeding, infectious inflammation, perforation, obstruction, or diarrhea greater than grade 1);
* NRS pain score ≥ 4 after standardized treatment with analgesics;
* Second primary malignancy within 5 years (except cured carcinoma in situ, basal cell, or squamous cell skin cancer; subjects with other previous tumors can be enrolled if there has been no recurrence within 5 years);
* Uncontrolled cardiovascular or cerebrovascular diseases with clinical symptoms, including but not limited to: ① NYHA class III or higher heart failure; ② unstable angina; ③ myocardial infarction or stroke within 6 months; ④ supraventricular or ventricular arrhythmias requiring treatment or intervention; ⑤ uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg despite optimal treatment);
* Known active hepatitis B subjects (HBsAg positive and HBV DNA ≥ 10³ copies or ≥ 1000 U/ml);
* Active infection or unexplained fever > 38.5°C during the screening period or on the day of administration (subjects with fever caused by tumors can be enrolled as judged by the investigator), which, in the investigator's judgment, would affect the subject's participation in this trial or interfere with the evaluation of efficacy;
* Known allergy to any components of irinotecan hydrochloride liposome, other liposomes, oxaliplatin, 5-FU, LV, or S-1;
* Pregnant or breastfeeding women;
* Women of childbearing potential with a positive blood (urine) pregnancy test during the screening period (both male and female subjects should use reliable contraception during the trial and for 3 months after the last dose to prevent pregnancy);
* Subjects with other medical or social issues that, in the investigator's judgment, might affect their ability to sign informed consent, participation in the trial, or interpretation of the trial results;
* Patients with an estimated survival time of ≤ 3 months are not included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From enrollment to the death from any cause, assessed up to 18 months

SECONDARY OUTCOMES:
Progression Free Survival | From enrollment to tumor progression or date of death from any cause, whichever came first, assessed up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No